CLINICAL TRIAL: NCT05711875
Title: The Effects of Using Virtual Reality Glasses on Anxiety, Stress, and Fetal Well-Being During the Non-Stress Test
Brief Title: The Effects of Using Virtual Reality Glasses During the Non-Stress Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Collaborators: İnönü University (Unknown)
Responsible Party: Principal Investigator, Mevhibe Coban, PhD student, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/2302
Record Dates: First submitted 2023-01-26; First posted 2023-02-03 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-01

CONDITIONS: Pregnancy Related
Keywords: Anxiety; non-stress test; stress; virtual glasses
MeSH Terms: conditions — Anxiety Disorders | interventions — Eyeglasses

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized controlled trial conducted with experimental and control groups (71 experimental group, 71 control group).
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Glasses (Experimental): Virtual Reality (VR) glasses applied group
  Interventions: Other: Virtual Reality (VR) glasses
- Standard of care (No Intervention): group without Virtual Reality (VR) glasses

INTERVENTIONS:
Other: Virtual Reality (VR) glasses — During the Non Stress Test (NST), the pregnant women in the experimental group watched a video of nature scenery with Virtual Reality (VR) glasses for 10 minutes
  Arms: Virtual Reality Glasses

SUMMARY:
The aim of this study to determine the effect of virtual reality glasses use on anxiety, stress and fetal well-being during the non-stress test. Personal information form was used as data collection form, Revised Prenatal Distress Questionnaire (NUPDQ-17 Item Version) was used to assess distress, State-Trait Anxiety Inventory (STAI) was used to assessanxiety.

DETAILED DESCRIPTION:
Material and Method

This research was conducted between between October 2021 and February 2022 in Fethi Sekin City Hospital. When power analysis was performed, the sample size was calculated to be at least 71 women for each group (71 experiments, 71 controls). During the NST procedures, VR glasses were given to the participants in the experimental group by the researcher for the intervention. Data collection form for experimental and control groups before the NST procedures; Revised Prenatal Distress Questionnaire (NUPDQ-17 Item Version) and State-Trait Anxiety Inventory (STAI) were applied two times before and after NST procedure. After the NST procedures, both groups were re-administered. Descriptive statistics and independent t-test were used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* not carrying any risk factors (e.g., preeclampsia, intrauterine growth retardation (IUGR), premature rupture of membranes, gestational diabetes)
* having a singleton pregnancy and no vision problems
* No uterine contraction on the tracing paper at the end of NST
* having eaten at least two hours before NST
* not smoking or drinking alcoholic beverages at least two hours before NST
* having a systolic blood pressure value in the range of 90-140 mmHg and a diastolic blood pressure value in the range of 60-90 mm/Hg
* not having any problems related to the health of the fetus (such as fetal anomaly, intrauterine growth retardation)
* having no communication barriers.

Exclusion Criteria:

* presence of fetal distress and emergency intervention planned by the physician
* uterine contraction as a result of NST

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Anxiety scores | NST involves 20 minutes of monitoring the fetal heart rate (FHR)
  StateTrait Anxiety Scale (STAI The highest score from the scale is 80, the lowest score is 20. Higher STAI-I scores indicate higher state anxiety levels
Distress scores | NST involves 20 minutes of monitoring the fetal heart rate (FHR)
  Revised Prenatal Distress Questionnaire (NUPDQ-17 Item Version): The highest score from the scale is 34, the lowest score is 0. Higher scores indicate higher levels of perceived prenatal distress in the respondent

SECONDARY OUTCOMES:
Fetal Well-Being scores | NST involves 20 minutes of monitoring the fetal heart rate (FHR)
  NST Registration Form: In the interpretations, the baseline FHR was accepted as 110-160 bpm, variability in a reactive NST was accepted as an FHR of 6-25 bpm, and acceleration was accepted as an elevation in the baseline FHR by at least 15 bpm for at least 15 s. Additionally, deceleration was accepted as a 15-20 bpm drop in comparison to the baseline FHR, and a reactive NST was defined as a result where two or more accelerations peaked at least 15 bpm above the baseline point, each acceleration lasted 15 s or longer, and all these conditions were met within 20 min from the start of the test. A nonreactive NST was defined as the absence of at least two accelerations lasting at least 15 s on the NST tracing paper within 20 min from the start of the test

CONTACTS AND LOCATIONS:
Overall Officials: ESRA GÜNEY, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
research results will be shared.

REFERENCES:
- [Result] Sridhar A, Shiliang Z, Woodson R, Kwan L. Non-pharmacological anxiety reduction with immersive virtual reality for first-trimester dilation and curettage: a pilot study. Eur J Contracept Reprod Health Care. 2020 Dec;25(6):480-483. doi: 10.1080/13625187.2020.1836146. PMID 33140989
- See also: Reference link — https://pubmed.ncbi.nlm.nih.gov/33140989/
- Available data/document: Informed Consent Form: Sridhar A, Shiliang Z, Woodson — https://pubmed.ncbi.nlm.nih.gov/33140989/ — web site is provided